CLINICAL TRIAL: NCT00005906
Title: Treatment With Octreotide in Patients With Lymphangioleiomyomatosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Joel Moss, M.D./National Heart, Lung and Blood Institute, National Institutes of Health
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 000147; 00-H-0147 (Other: NHLBI)
Record Dates: First submitted 2000-06-09; First posted 2000-06-12 (Estimated); Results first posted 2010-04-30 (Estimated); Last update posted 2010-04-30 (Estimated); Status verified 2010-04

CONDITIONS: Lymphangioleiomyomatosis; Lymphangiomyomas; Pleural Effusions; Ascites
Keywords: Chylous Ascites; Chylous Pleural Effusion; Inhibitory Effects; Lymphangioleiomyoma; Somatostatin; Lymphangioleiomyomatosis (LAM)
MeSH Terms: conditions — Lymphangioleiomyomatosis; Lymphangiomyoma; Pleural Effusion; Ascites; Chylous Ascites; Chylothorax | interventions — Octreotide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Octreotide (Experimental): Patients with lymphangioleiomyomatosis and lymphatic tumors, ascites or pleural effusions who are symptomatic will receive subcutaneous injections of octreotide starting at a dose of 100 micrograms per day. Doses will be gradually increased to a maximum of 800 micrograms per day, two months after enrollment, if there is no response to lower doses.
  Interventions: Drug: Octreotide

INTERVENTIONS:
Drug: Octreotide — Treatment with octreotide starts at a dose of 50 micrograms(ug) twice a day which is increased to 100 ug twice a day after two weeks and to 200 ug twice a day two weeks later. After two months, if there is no response the dose shall be increased to 400 ug twice a day.

SUMMARY:
Lymphangioleiomyomatosis (LAM), a disease primarily of women of child-bearing age, is characterized by cystic lung disease and abdominal tumors (e.g., angiomyolipomas). Within the LAM patient population is a subset of patients who develop chylous effusions and lymphangioleiomyomas. Treatment of many of these symptoms has been ineffective. Previous studies with somatostatin and octreotide in other clinical settings have shown reduction in chylous effusions. This study assesses the effectiveness of octreotide in symptomatic patients with LAM, lymphangioleiomyomas and/or chylous effusions/ascites, peripheral lymphedema and chyluria.

DETAILED DESCRIPTION:
Lymphangioleiomyomatosis (LAM), a disease primarily of women of child-bearing age, is characterized by cystic lung disease and abdominal tumors (e.g., angiomyolipomas). Within the LAM patient population is a subset of patients who develop chylous ascites, chylous pleural effusions, chyluria, peripheral lymphedema, and/or lymphangioleiomyomas. Lymphangioleiomyomas are believed to result from a proliferation of abnormal smooth muscle cells within the lymphatic system, which appears to obstruct fluid outflow, leading to fluid accumulation and an increase in size. The lymphangioleiomyomas may occur anywhere along the axial lymphatic chain. In patients with LAM, they occur most frequently in the thorax, abdomen and pelvis and may give rise to a myriad of symptoms (e.g., paresthesias, palpitations, peripheral edema). In some patients, treatment of many of these symptoms, i.e., elevation of lower extremities, paracentesis, thoracentesis, diuretics, and/or surgery, has been ineffective. Previous studies with somatostatin and octreotide in other clinical settings (e.g., traumatic damage to the lymphatics) have shown a successful reduction in chylous effusions, chyluria, ascites, and peripheral lymphedema, when other therapies were less effective. This study will assess the effectiveness of octreotide in symptomatic patients with LAM, lymphangioleiomyomas and/or chylous effusions/ascites, peripheral lymphedema and chyluria. The dose of octreotide starts at 50 micrograms (ug) by the subcutaneous route twice a day. After two weeks the dose will be increased to 200 ug per day and two weeks later to 400 ug/day. Maximal dose is 400 ug twice a day.

ELIGIBILITY:
* INCLUSION CRITERIA:

Patients enrolled in the lymphangioleiomyomatosis natural history protocol who have symptoms associated with one of the following:

1. lymphangioleiomyomas
2. chylous pleural effusions
3. peripheral lymph-edema
4. chyloptysis
5. protein-losing enteropathy
6. chyluria

Patients will be included in this protocol if symptoms are attributed to the above processes. Patients with malabsorption disorders, diabetes, hypo/hyperthyroidism, or other endocrine-related disorders will be included if justified clinically based on severity of symptoms.

EXCLUSION CRITERIA:

1. Hypersensitivity to somatostatin, octreotide or its analogues
2. Patients with hepatitis B, hepatitis C, or other clinically significant liver diseases
3. Transplant patients
4. Pregnant women or women who are beast-feeding
5. Patient or another responsible party is unable to give the subcutaneous injection
6. Patient unwilling to be followed per the guidelines set forth
7. Patients with decreased renal function (creatinine greater than 1.5)
8. Patients with HIV infection
9. Immunosuppressed patients

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2000-06; Primary Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Ulibarri JI, Sanz Y, Fuentes C, Mancha A, Aramendia M, Sanchez S. Reduction of lymphorrhagia from ruptured thoracic duct by somatostatin. Lancet. 1990 Jul 28;336(8709):258. doi: 10.1016/0140-6736(90)91793-a. No abstract available. PMID 1973814

RESULTS

PARTICIPANT FLOW:
Groups:
- Octreotide: Patients with lymphangioleiomyomatosis and lymphatic tumors causing chylous effusions and abdominal pain
Period: Overall Study
Arm/Group | Octreotide
Started | 4
Completed | 1
Not Completed | 3
Not completed — Lack of Efficacy | 3

BASELINE CHARACTERISTICS:
Arm/Group | Octreotide
Number analyzed (Participants) | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 43 (5.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 4

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a Reduction in Total Tumor Volume of at Least 20%.
Description: Octreotide treatment will be considered successful if the patient receiving treatment for six months shows a reduction in total tumor mass/ fluid collection or reaccumulation of at least 20%.
Time Frame: Six months
Measure: Number; unit: Participants
Arm/Group | Octreotide
Number analyzed (Participants) | 4
Participants | 0 (5)

2. Primary Outcome: Number of Participants With a Reduction of Pain/Symptoms as Measured by a Simple Numeric Symptom Distress Scale (NDS) to Rate the Severity of Individual Symptoms.
Description: Octreotide treatment will be considered successful if the reported pain/symptom score is reduced by at least 2 levels at termination of treatment.
  A simple visual numeric distress scale ranging from zero to 10 will be employed to rate the severity of individual symptoms. The best score is zero, which means absence of symptoms and the maximal is 10, meaning that the symptoms are very severe.
Time Frame: Six months
Population: Four patients with lymphangioleiomyomatosis and lymphangioleiomyomas and chylous effusions treated with octreotide injections by the subcutaneous route to determine whether the size of the tumors and effusions decrease with the therapy
Measure: Number; unit: Participants
Arm/Group | Octreotide
Number analyzed (Participants) | 4
Participants | 1 (5)

3. Secondary Outcome: Number of Participants With Liver Function Abnormalities
Description: One or more abnormality of the following liver function tests:
  1. Alkaline phosphatase above 116 i.u.
  2. SGPT above 41 i.u.
  3. SGOT from 34 i.u.
  4. Total bilirubin above 1.0 mg/dl
Time Frame: Six months
Measure: Number; unit: Participants
Arm/Group | Octreotide
Number analyzed (Participants) | 4
Participants | 1

ADVERSE EVENTS:
Arm/Group | Octreotide
Serious Adverse Events (participants affected / at risk) | 1/4
Other Adverse Events (participants affected / at risk) | 1/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Octreotide (N=4)
Gastrointestinal disorders (Hepatobiliary disorders) | 1 (1) — On September 2000 the patient referred right upper quadrant abdominal pain. An abdominal ultrasound showed gallbladder sludge. Octreotide was discontinued. In December, an ultrasound showed gallstones. In February 2001 she had a cholecystectomy.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Octreotide (N=4)
Liver function abnormalities (Gastrointestinal disorders) | 1 (1) — Mild elevation of liver function tests.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No